CLINICAL TRIAL: NCT03770832
Title: Wearable Sensors and Video Recording for Children (Birth to 24 Months) to Monitor Motor Development
Brief Title: Wearable Sensors and Video Recordings to Monitor Motor Development
Status: Active, not recruiting | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); Northwestern University (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Other Study IDs: SX04202018
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Motor Delay; Neurodevelopmental Disorders; Developmental Disability
Keywords: Early Detection; Wearable Sensors; Computer Vision
MeSH Terms: conditions — Psychomotor Disorders; Neurodevelopmental Disorders; Developmental Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants at Risk for Atypical Motor Development (high-risk)
- Infants Expected to Have Typical Motor Development (low-risk)

SUMMARY:
The objective of this study is to develop an automated, precise, quantitative assay for detecting atypical motor behavior and development in infants using data from wearable sensors and video recordings.

ELIGIBILITY:
Inclusion Criteria:

* Individuals identified as potentially at risk of abnormal motor development due to a risk factor (for example, prematurity, neonatal hypoxic ischemic encephalopathy, or neonatal stroke) OR control individuals for whom normal motor development is expected.
* Age: < 24 months of age
* Legal guardian able and willing to give written consent and comply with study procedures.
* In case of multiple pregnancies, only one child selected at random will participate in the research activities. Study staff will have no influence over the selection, besides any known medical condition automatically excluding the baby as listed in our exclusion criteria.

Exclusion Criteria:

* Any open wound or skin breakdown on the limbs or upper torso.
* Missing or incomplete limbs (such as from amputation or congenital limb defects)
* Legal guardian unable to give written consent and comply with study procedures.

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Individuals at high risk of developing motor delays <24 months of age along with infants at low risk of developing motor delays.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Three month clinical score estimation | 3 months
  Error between true clinical test scores and scores estimated from sensor and video data, assessed at the 3 month time-point.
Six month clinical score estimation | 6 months
  Error between true clinical test scores and scores estimated from sensor and video data, assessed at 6 month time-point.
Prediction of neuromotor outcome using sensor and video data from 3 month time-point | 3 months
  Sensitivity and specificity of algorithm (trained on sensor and video data from the 3 month time-point) to predict neuromotor outcome at final study visit (as measured by the Peabody Developmental Motor Scales, second edition [PDMS-2])
Prediction of neuromotor outcome using sensor and video data from 6 month time-point | 6 months
  Sensitivity and specificity of algorithm (trained on sensor and video data from the 6 month time-point) to predict neuromotor outcome at final study visit (as measured by the Peabody Developmental Motor Scales, second edition [PDMS-2])

SECONDARY OUTCOMES:
Prediction of neuromotor outcome using General Movements Assessment (GMA) scores | 1-2 weeks, 1 month, 3 months
  Sensitivity and specificity of GMA scores (taken at 1-2 weeks, 1 month, 3 months) to predict neuromotor outcome at final study visit (as measured by the Peabody Developmental Motor Scales, second edition [PDMS-2]). The GMA is an observational exam where an infant's spontaneous movements are scored as atypical or normal for their age.
Prediction of neuromotor outcome using Alberta Infant Motor Scale (AIMS) scores | 6 months, 9 months, 1 year
  Sensitivity and specificity of AIMS scores (taken at 6 months, 9 months, 1 year) to predict neuromotor outcome at final study visit (as measured by the Peabody Developmental Motor Scales, second edition [PDMS-2]). The AIMS is a norm-referenced observational assessment with a minimum score of 0 and a maximum score of 58. Higher scores indicate better motor performance on the assessment.
Prediction of neuromotor outcome using Hammersmith Infant Neurological Examination (HINE) scores | 6 months, 9 months, 1 year
  Sensitivity and specificity of HINE scores (taken at 6 months, 9 months, 1 year) to predict neuromotor outcome at final study visit (as measured by the Peabody Developmental Motor Scales, second edition [PDMS-2]). The HINE is a neurological exam with a minimum score of 0 and a maximum score of 78. Higher scores indicate better performance on the assessment.
Prediction of neuromotor outcome using Test of Infant Motor Performance (TIMP) scores | 1-2 weeks, 1 month, 3 months
  Sensitivity and specificity of TIMP scores (taken at 1-2 weeks, 1 month, 3 months) to predict neuromotor outcome at final study visit (as measured by the Peabody Developmental Motor Scales, second edition [PDMS-2]).
Clinical score estimation | 1-2 weeks, 1 month, 9 months, 1 year, 2 years
  Error between true clinical test scores and scores estimated from sensor and video data, assessed at each remaining time-point.
Prediction of neuromotor outcome at 2 years using sensor and video data from the remaining time-points | 1-2 weeks, 1 month, 9 months, 1 year, 2 years
  Sensitivity and specificity of algorithm (trained on sensor and video data from the remaining time-points) to predict neuromotor outcome at 2 years (as measured by the Peabody Developmental Motor Scales, second edition [PDMS-2])

OTHER OUTCOMES:
Prediction of neuromotor outcome using NICU Network Neurobehavioral Scale (NNNS) scores | 1 month
  Sensitivity and specificity of NNNS scores (taken at 1 month) to predict neuromotor outcome at final study visit (as measured by the Peabody Developmental Motor Scales, second edition [PDMS-2])

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (2):
- United States (2):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois